CLINICAL TRIAL: NCT03698058
Title: Real-World Effectiveness Study of A2 Growing Up Milk (GUM) Among Young and Pre-School Age Toddlers in China
Brief Title: A2 GUM Post-Market Effectiveness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18.14.INF
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Protein Intolerance
Keywords: Nutrition; Toddlers; A2; B-casein; Gut comfort; Growing up milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A2 Growing Up Milk (Experimental)
  Interventions: Dietary Supplement: Toddler milk
- Traditional non-A2 milk (No Intervention)
- Other Growing Up Milk (Active Comparator)
  Interventions: Dietary Supplement: Toddler milk

INTERVENTIONS:
Dietary Supplement: Toddler milk — Commercially available toddler milk
  Arms: A2 Growing Up Milk; Other Growing Up Milk

SUMMARY:
This is a post-market, real-life effectiveness study of A2 growing up milk on toddlers' gut comfort.

DETAILED DESCRIPTION:
This post-market study primarily aims to assess the real-life effectiveness of a newly-launched A2 milk on toddlers' gut comfort via evaluating individual GI symptoms and GI-related behaviors compared with other milk products and milk alternatives.

ELIGIBILITY:
Inclusion Criteria:

* Having obtained his / her parents' (or his or her legally accepted guardian written informed consent and having evidence of personally signed and dated informed consent document indicating that the child's parent(s) / legal guardian has been informed of all pertinent aspects of the study.
* Children 12 - 36 months of age at enrolment.
* Children who have been born full-term (≥ 37 completed weeks of gestation) and having a birth weight ≥ 2.5 kg and ≤ 4.5 kg.
* Children who are habitually consuming some cow's milk, other traditional milks (including non-A2 GUMs, kids' milk, white milk, flavored milk) and/or dairy or non-dairy alternative milks (such as those sourced from goats, sheep, soy, rice, coconut, and nut).
* Child's parent(s) / guardian is of legal age of consent, has sufficient command of Chinese (Mandarin) language to complete the informed consent and other study documents, is willing and able to fulfill the requirements of the study protocol.

Exclusion Criteria:

* Chronic infectious, metabolic, genetic illness or other disease including any condition that impacts feeding or may impact outcome measures.
* Known and diagnosed cow's milk protein allergy.
* Children currently using or having ever used specialty infant formula and/or GUMs such as hypoallergenic (HA), lactose-free, or anti-regurgitation formulas.
* Children who have known cognitive and developmental disorders.

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 387 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Overall digestive comfort | Baseline to Study Day 14
  Toddler Gut Comfort score from parent-reported questionnaire (sub-scale range from 1 to 6, 10 sub-scales, total scores range from 10-60).

SECONDARY OUTCOMES:
Stool frequency | Baseline, Study Day 7, Study Day 14
  Stool frequency reported by parents in 3-Day GI Symptoms Diary
Stool consistency | Baseline, Study Day 7, Study Day 14
  Stool consistency score reported by parents in 3-Day GI Symptoms Diary
Consumption of other milk products | Baseline, Study Day 7, Study Day 14
  Reported by parents on 3 consecutive days on Milk Intake Diary
Child weight | Baseline, Study Day 7, Study Day 14
  Weight as measured by study staff in health clinic
Child height | Baseline, Study Day 7, Study Day 14
  Weight as measured by study staff in health clinic
Child head circumference | Baseline, Study Day 7, Study Day 14
  Head circumference as measured by study staff in health clinic
Adverse events | Baseline to Study Day 14
  All adverse events reported by parents and confirmed by study investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Reproductive and Child Health, Peking University, Beijing, China

IPD SHARING:
Plan to Share IPD: No